CLINICAL TRIAL: NCT06955065
Title: Effects of Battle Rope Training Program On Bocce Throwing In Young Adaptive Bocce Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/KHADIJA KIRAN
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Special Senses Disorders
Keywords: Battle training; bocce throwing; adaptive sports; upper body strength; coordination
MeSH Terms: conditions — Sensation Disorders

STUDY DESIGN:
Intervention Model Description: This study will be randomized controlled trial. It will include 18 young adaptive bocce players aged 10 to 18 years who meet the inclusion criteria, such as having a physical disability that qualifies them for adaptive sports, being able to understand and follow instruction, and having no recent injuries or surgeries that would contraindicated exercise.
  Participant will be randomly assigned to either the experimental group, which will undergo a structured battle rope training or the control group which will continue with their regular bocce training regimen. The battle rope training program will be designed to enhance upper body strength, endurance, and coordination and will be conducted three times a week for 8 weeks.pre and post intervention will include
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Battle Rope Training (Experimental): Participants in the experimental group will undergo a structured battle rope training program. Total duration is 8 weeks and perform 3 session per week, for 30 seconds with 10 second rest period. The program will progressively increase in intensity and complexity to challenge participants' upper body strength, coordination, and endurance, intensity and complexity to challenge participants' upper body strength, coordination and endurance
  Interventions: Other: battle rope training
- Bocce Throwing (Active Comparator): Participants in the control group will engage in regular bocce training sessions as per their usual routine. These sessions will focus on standard bocce drills and techniques without additional battle rope exercise .A warm up activity used in every training session and a proper warm-up should include Aerobic activity and Dynamic stretching for 15 to 20 repetitions of each exercise.
  Interventions: Other: Bocce Throwing

INTERVENTIONS:
Other: battle rope training — Battle rope training is a dynamic, high-intensity exercise involving heavy ropes to improve strength, endurance, and coordination. It primarily targets the upper body, including the shoulders, arms, and core, through rhythmic, wave-like movements. This training is adaptable and effective for enhancing functional fitness in both general and adaptive athletes.
  Arms: Battle Rope Training
Other: Bocce Throwing — Participants in the control group will engage in regular bocce training sessions as per their usual routine. These sessions will focus on standard bocce drills and techniques without additional battle rope exercise. A warm- up activity used in every training session and a proper warm-up should include Aerobic activity and Dynamic stretching . 15 to 20 repetitions of each exercise.
  Arms: Bocce Throwing

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of battle rope training in enhancing athletic performance among young adaptive bocce players aged 10 to 18 years. A total of 18 participants with physical disabilities qualifying them for adaptive sports, capable of following instructions and without recent injuries or surgeries, will be randomly assigned to either an experimental group undergoing structured battle rope training or a control group continuing regular bocce training. The 8-week intervention, conducted three times per week, focuses on improving upper body strength, endurance, and coordination. Pre- and post-intervention assessments will include bocce throwing accuracy and distance, grip strength, number of rope slams in a set time, and shoulder endurance, with a dynamometer used to measure strength metrics. Data will be analyzed using SPSS version 23 to determine the impact of battle rope training on performance and fitness in adaptive sports

DETAILED DESCRIPTION:
Adaptive sports offer individuals with physical disabilities opportunities for competitive and recreational engagement, promoting physical fitness, social interaction and overall wellbeing. Among these sport, bocce stands out as a precision ball sport similar to bowling, requiring players to develop fine motor skills, coordination and upper body strength for effective throwing. Enhancing upper body strength, coordination and endurance is crucial for improving performance in bocce especially for adaptive players who may have physical limitation. This study aims to provide evidence for the incorporation of battle rope training into the training routines of young adaptive bocce players. Positive results could lead of the broader adoption of battle rope exercise, thereby enhancing athletic performance and physical fitness in adaptive sports. This study will be randomized controlled trial. It will include 18 young adaptive bocce players aged 10 to 18 years who meet the inclusion criteria, such as having a physical disability that qualifies them for adaptive sports, being able to understand and follow instruction, and having no recent injuries or surgeries that would contraindicated exercise.

Participant will be randomly assigned to either the experimental group, which will undergo a structured battle rope training or the control group which will continue with their regular bocce training regimen. The battle rope training program will be designed to enhance upper body strength, endurance, and coordination and will be conducted three times a week for 8 weeks pre and post intervention will include measurement of bocce throwing performance, especially accuracy and distance, as well as upper body strength and endurance tests, such as grip strength, the number of rope slams performed in a given time and shoulder endurance tests. Dynamometer is used to measure weight and pull forces.

Data will be analyzed through SPSS version 23

ELIGIBILITY:
Inclusion Criteria:

* Young adaptive bocce players aged between 10 to 16 years.
* Diagnosed with a disability that qualifies them for adaptive sports participation.
* Ability to comprehend and follow instructions related to the study protocol

Exclusion Criteria:

* Recent injuries or surgeries that affect upper body function or overall physical activity.
* Non-compliance with the study protocol or inability to participate regularly in training sessions
* Severe cognitive impairments that hinder understanding of instructions and participation in assessment

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Bocce Throwing Performance | baseline,6th week
  Bocce throwing performance refers to a player's ability to accurately and consistently throw balls close to the target assessed by precision, distance control, and consistency. Performance measures are considered valid as they reflect actual game skills and reliable due to consistent outcomes under similar conditions.
Grip Strength measurement bt Dynamometer | baseline,6th week
  Calibrated dynamometer is used to measure the grip strength. participant s elbow should be at 90-degree angle and positioned at the side of their body. ensure that hand is neutral position and thumb facing up. Instruct the participant to squeeze the dynamometer handle about 3 to 5 seconds.
  Repeat the measurement three times for each hand, with rest period of 30 seconds.
Rope slams in 30 seconds | baseline,6th week
  Ensure the battle rope is 20m long 1.5cm in diameter and securely anchored. The participant stand with feet shoulder-width apart, holding one end of the rope in each hand with fully extended arms in front of body ,slightly bend knees and straight back .On commands , go the the participant will start performing alternating rope slams as quickly and forcefully as possible .Count the number of complete slams within 30 seconds period. Test -retest reliability of upper body was reported by ICC within day sessions. The within day ICC for upper body power was 0.890.
upper Limb Functional Index | baseline,6th week
  upper Limb Functional Index: The upper limb functional index is a tool to assess functional limitation in the upper limb, particularly the shoulder ,elbow, forearm and hand.it consist of a questionnaire that evaluate the difficulty individuals have with various activities of daily living due to upper limb impairment . Test-retest reliability and consistency of Upper limb functional index was good internal consistency was within range of 0.75 to 0.95. An ICC value ≥ 0.70 would support the test-retest reliability of the Upper limb functional test

CONTACTS AND LOCATIONS:
Overall Officials: khadija kiran, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Insititute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen WH, Yang WW, Lee YH, Wu HJ, Huang CF, Liu C. Acute Effects of Battle Rope Exercise on Performance, Blood Lactate Levels, Perceived Exertion, and Muscle Soreness in Collegiate Basketball Players. J Strength Cond Res. 2020 Oct;34(10):2857-2866. doi: 10.1519/JSC.0000000000002661. PMID 30024481